CLINICAL TRIAL: NCT06144606
Title: Phase 2 Study of KTE-X19 in Minimal Residual Disease (MRD) Positive B-Cell Acute Lymphoblastic Leukemia (B-ALL)
Brief Title: Study of KTE-X19 in Minimal Residual Disease (MRD) Positive B-Cell Acute Lymphoblastic Leukemia (B-ALL)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-22286
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: B-Cell Lymphoblastic Leukemia; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — brexucabtagene autoleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous CAR T-cell immunotherapy (Experimental): Tecartus will be delivered at a target dose of 1x106 cells / kg. For those >100 kg, a flat dose of 1 x108 cells will be used. Tecartus will be administered on day 0, following 1 day of rest from conditioning chemotherapy.
  Interventions: Drug: Tecartus

INTERVENTIONS:
Drug: Tecartus — Tecartus is a CD19 directed CAR T-cell therapy that utilizes CD28 costimulatory and CD3 zeta stimulatory domains. Tecartus is manufactured from purified autologous T-cells via retroviral transduction with a median time to product release of 13 days.
  Other Names: Brexucabtagene autoleucel; KTE-X19

SUMMARY:
This is a Phase 2 Study is to determine the efficacy and safety rate of B-Cell Acute Lymphoblastic Leukemia (B-ALL) participants in remission with minimal residual disease (MRD) after KTE-X19 CAR T-cell therapy

ELIGIBILITY:
Inclusion Criteria:

* Must be an adult 18 years of age or older.
* Pathologically confirmed CD19 positive B-cell acute lymphoblastic leukemia.
* Treatment and full recovery from induction chemotherapy, with following exceptions:

A. Vincristine associated grade 1 peripheral neuropathy B. Steroid/asparaginase associated diabetes and/or hypertension C. Inotuzumab/chemotherapy associated cytopenias

* Patients must be in a complete remission with Minimal Residual Disease (MRD) following an induction regimen. MRD is defined herein as a bone marrow biopsy with fewer than 5% lymphoblasts. Complete remission implies the resolution of any extramedullary and/or Central Nervous Syndrome (CNS)-2-3/parenchymal disease.
* Be willing and able to provide written informed consent/assent for the trial.
* Able to adhere to the study visit schedule and other protocol requirements.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Adequate renal, hepatic, pulmonary, cardiac function.
* Adequate hematopoietic reserve.
* Females of childbearing potential (FCBP) must have a negative serum pregnancy test at screening. A FCBP is considered when a sexually mature female:

  1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months.
* Subjects of both genders of child-bearing potential must be willing to practice birth control from the time of consent through 6 months after the completion of KTE-X19 infusion.

Exclusion Criteria:

* Diagnosis of L3 type Burkitt's lymphoma, Mixed-Lineage Leukemia (MLL) rearranged leukemia, biphenotypic leukemia, mixed phenotype acute leukemia, blast phase of chronic myeloid leukemia, or stem-cell leukemia.
* Any active infection requiring systemic therapy, including HIV, Hepatitis B, and/or Hepatitis C.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator (including but not limited to unstable angina, pre-existing liver disease, recurrent pancreatitis, uncontrolled diabetes, hypertriglyceridemia, pulmonary hypertension, or severe Congestive Heart Failure (CHF).
* Recurrent thrombosis, or non-central venous catheter associated thrombosis within 3 months prior to enrollment.
* History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment.
* History or presence of any CNS disorder such as a seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, any autoimmune disease with CNS involvement, posterior reversible encephalopathy syndrome (PRES), or cerebral edema.
* Active CNS/leptomeningeal leukemia.
* Severe comorbid conditions for which life expectancy would be <6 months.
* Patients with active (uncontrolled, metastatic) second malignancies are excluded.
* History of concomitant genetic syndrome associated with bone marrow failure such as Fanconi anemia, Kostmann syndrome, Shwachman-Diamond syndrome.
* Primary immunodeficiency or history of autoimmune disease (Crohns, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years.
* Corticosteroid therapy at a pharmacologic dose (> 5 mg/day of prednisone or equivalent doses of other corticosteroids) and other immunosuppressive drugs must be avoided for 7 days prior to enrollment.
* Presence of any indwelling line or drain (percutaneous nephrostomy tube, indwelling Foley catheter, biliary drain, or pleural/peritoneal/pericardial catheter). Ommaya reservoirs and dedicated central venous access catheters such as a Port-a-Cath or Hickman catheter are permitted.
* Live vaccine ≤ 4 weeks prior to enrollment.
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 3 months after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-26 (Actual); Primary Completion 2028-11-15 (Estimated); Study Completion 2028-11-15 (Estimated)

PRIMARY OUTCOMES:
Relapse Free Survival (RFS) | Up to 5 years
  The primary endpoint is RFS, defined as the time from KTE-X19 infusion until clinical relapse or death from any cause. Patients proceeding to subsequent anti-cancer therapy, inclusive of allogeneic transplantation, without relapse will be censored in this analysis. Surviving patients not meeting criteria for relapse by the analysis data cutoff date will be censored at their last evaluable disease assessment date.

SECONDARY OUTCOMES:
Molecular Response Rate | Up to 5 years
  Measured as converting to a complete molecular remission following CAR T-cell immunotherapy. Molecular remission is defined as having fewer than 0.0001% clonotype sequences per one million nucleated cells.
Clinical Relapse Rate | Up to 5 years
  Measured as >5% lymphoblasts in the bone marrow and/or the emergence of extramedullary leukemia.
Molecular Relapse Rate | Up to 5 years
  Measured as achieving complete molecular remission at day 28 and followed until 5 years from infusion or the emergence of detectable disease.
  Molecular remission is defined as having fewer than 0.0001% clonotype sequences per one million nucleated cells.
Duration of Response (DOR) | Up to 5 years
  Measured as time from enrollment until clinical relapse or death. In the case of death without documented relapse, patients will be censored.
Molecular Relapse Free Survival (MRFS) | Up to 5 years
  Measured by complete molecular remission at day 28 and followed until 5 years from infusion or the emergence of detectable disease.
  Molecular remission is defined as having fewer than 0.0001% clonotype sequences per one million nucleated cells.
Overall Survival | Up to 5 years
  Measured as time from date of enrollment to date of death from any cause.
Rate of Cytokine Release Syndrome (CRS) | Up to 5 years
  Participants rate of developing Cytokine Release Syndrome (CRS)
Rate of Immune effector cell-associated neurotoxicity syndrome (ICANS) | Up to 5 years
  Participants rate of developing Immune effector cell-associated neurotoxicity syndrome (ICANS).

CONTACTS AND LOCATIONS:
Overall Officials: Bijal D. Shah, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States